CLINICAL TRIAL: NCT06638333
Title: Prevalence and Serotype Distribution of Streptococcus Pneumoniae in Healthy Vietnamese Children From 6 Months to 5 Years Old
Status: Active, not recruiting | Type: Observational
Sponsor: Tam Anh Research Institute (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Other Study IDs: TA0002
Record Dates: First submitted 2024-10-09; First posted 2024-10-15 (Actual); Last update posted 2025-04-13 (Actual); Status verified 2025-03

CONDITIONS: Streptococcus Pneumonia
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Observational Model: Ecologic or Community | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Nasopharyngeal sample will be put in retention without analysis of human DNA
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- Children between 6 months and 5 years

SUMMARY:
This observational study is designed as a cross-sectional survey of children from 6 months and 5 years old who visit the Vietnam Vaccination Center (VNVC) system in Hanoi, Danang and Ho Chi Minh City for vaccination services.

After getting the informed consent form from a parent/guardian for their child(s) to participate in the study, nasopharyngeal swab sample will be taken. His/her guardian will be interviewed face-to-face with information related to epidemiological characteristics, nutritional status, child's birth history, hospitalization history, vaccination history, recent antibiotic usage, breastfeeding time, and environmental and lifestyle factors.

The goal is to document the burden and risk factors of pneumococcal infections in the community of healthy Vietnamese children. The main questions it aims to answer are:

* What is the prevalence of pneumococcus in healthy children?
* What is the distribution of pneumococcus serotypes in the community of healthy Vietnamese children?
* What are risk factors of pneumococcus infection in the community of healthy Vietnamese children?

ELIGIBILITY:
Inclusion Criteria:

* Children between 6 months and 5 years

Exclusion Criteria:

* Children with chronic diseases (including immunologic diseases, neoplastic disorders, renal, cardiac, hepatic, or hematologic diseases, broncho dysplasia, Down syndrome, chronic otitis media with effusion)
* Children with acute/chronic upper or lower respiratory tract infection
* Children have used antibiotics within 1 week prior to entering the study

Ages: 6 Months to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children from 6 months and 5 years old who visit the Vietnam Vaccination Center (VNVC) system in Hanoi, Danang and Ho Chi Minh city for vaccination services
Sampling Method: Non-Probability Sample
Enrollment: 800 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-06-30 (Estimated); Study Completion 2025-06-30 (Estimated)

PRIMARY OUTCOMES:
Prevalence of pneumococcal carriage in the nasopharynx in children from 6 months to 5 years old in the Vietnamese community | Day 0 after recruitment
  Pneumococcal prevalence in children by age group, sex and geographical area
Serotype distribution of pneumococcal strains in Vietnamese children from 6 months to 5 years old in the community | Day 0 after recruitment
  The number of carrier individuals by serotype will be determined for age group, sex and geographical area

SECONDARY OUTCOMES:
Risk factors associated with pneumococcal carriage | Day 0 after recruitment
  Gender, age, urban vs rural setting, environmental, lifestyle factors and other factors will be analyzed.

CONTACTS AND LOCATIONS:
Locations (3):
- Vietnam (3):
  - VNVC Da Nang, Da Nang
  - VNVC Icon4 Cau Giay, Hanoi
  - VNVC Tan Phu, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: No